CLINICAL TRIAL: NCT04923932
Title: A Multi-center, Open-label, Phase II Clinical Trial to Evaluate the Efficacy, Safety and Tolerability of Savolitinib in Treating Gastric Cancer and Esophagogastric Junction Adenocarcinoma Patients With MET Gene Amplifications
Brief Title: Savolitinib for Treating Gastric Cancer and Esophagogastric Junction Adenocarcinoma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-504-00CH1
Record Dates: First submitted 2021-05-30; First posted 2021-06-11 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancer; Esophagogastric Junction Disorder
MeSH Terms: conditions — Stomach Neoplasms | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Intervention Model Description: locally advanced or metastatic Gastric Cancer and Esophagogastric junction adenocarcinoma Patients with MET gene amplifications with measurable lesions OR with no measurable lesions but have evaluable lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Savolitinib (Experimental): GC
  Interventions: Drug: Savolitinib

INTERVENTIONS:
Drug: Savolitinib — Patients meeting the study inclusion criteria will receive Savolitinib [Savolitinib 600 mg, po, once per day (QD) continuously in patients with baseline weight ≥50 kg, and Savolitinib 400 mg, po, QD in patients with baseline weight <50 kg] in 21 day treatment cycle, until disease progression, death, intolerable toxicity or other termination criteria as specified in the protocol, whichever occurs earliest.
  Other Names: hmpl-504

SUMMARY:
Treating Gastric Cancer and Esophagogastric junction adenocarcinoma Patients with MET gene amplifications with Savolitinib

DETAILED DESCRIPTION:
This is a single-arm, multi-cohort, multi-center, open-label, phase II clinical study. The objective is to evaluate the efficacy and safety of Savolitinib in the treatment of locally advanced or metastatic Gastric Cancer and Esophagogastric junction adenocarcinoma Patients with MET gene amplifications. The study involves a Screening Period, a Treatment Period and a Follow-up Period. It is planned that about 30 study sites will enroll 75 patients

ELIGIBILITY:
Inclusion Criteria:

1. Fully aware this study and signed the informed consent form in voluntary manner, and willing and able to comply with the study procedure;
2. Age ≥18 years;
3. Histologically diagnosed locally advanced or metastatic Gastric Cancer and Esophagogastric junction adenocarcinoma
4. MET gene amplifications
5. Cohort 1: Having measurable lesions (in accordance with RECIST 1.1 criteria); Cohort 2: having evaluable lesions
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2
7. Survival is expected to exceed 12 weeks;
8. Adequate functionality in bone marrow, liver, kidney
9. Able to take or swallow the drug orally.
10. Female patients of childbearing potential must agree to use effective contraceptive methods from screening period to 30 days after discontinuation of the study drug,The male patients whose sexual partners are women of childbearing age must use condom during sexual intercourse during the study and within 6 months after discontinuation of study drug;

Exclusion Criteria:

1. Currently having other malignant tumors, or having other infiltrating malignant tumors in the past 5 years. Stage I malignant tumor after radical treatment for at least 3 years, except those considered by investigators to have small possibility of recurrence. Patients with radically treated carcinoma in situ (non-infiltrating) and skin cancer other than malignant melanoma can be enrolled;
2. Having received antitumor therapy (including chemotherapy, hormone therapy, biotherapy, immunotherapy or traditional Chinese medicine for antitumor indication) within 3 weeks prior to the start of study treatment, or having received treatment with small molecular tyrosine kinase inhibitors (e.g., EGFR-TKI) within 2 weeks prior to the start of study treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) evaluated by the Independent Review Committee (IRC) (RECIST 1.1 criteria) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 42 months
  To evaluate the efficacy of Savolitinib in the treatment of locally advanced or metastatic Gastric Cancer and Esophagogastric junction adenocarcinoma Patients with MET gene amplifications

SECONDARY OUTCOMES:
Progression-free survival (PFS) (RECIST 1.1 criteria) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 42 months
  Efficacy of Savolitinib in the treatment of locally advanced or metastatic Gastric Cancer and Esophagogastric junction adenocarcinoma Patients with MET gene amplifications
incidence of various adverse events (AE) | through study completion, an average of 3.5 year
  To evaluate the safety and tolerability of Savolitinib in the treatment of locally advanced or metastatic Gastric Cancer and Esophagogastric junction adenocarcinoma Patients with MET gene amplifications

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hopspital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No